CLINICAL TRIAL: NCT05279625
Title: Effects of Exercise Interventions in Frail Middle-aged and Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-10-014BCF
Record Dates: First submitted 2022-01-25; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Frailty
Keywords: exercise; frailty; physical function; mental function; aged
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: a randomized, multi-arm parallel and controlled intervention study.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Interval exercise training (Experimental): Interval exercise training using either elastic band, dumbbells, treadmill, cycling for 6 months
  Interventions: Device: exercise training
- continuous exercise training (Experimental): continuous exercise training using either elastic band, dumbbells, treadmill, cycling for 6 months
  Interventions: Device: exercise training
- machine-assisted exercise training (Experimental): machine-assisted exercise training for 6 months
  Interventions: Device: exercise training
- traditional rehabilitation (Active Comparator): traditional rehabilitation for 6 months
  Interventions: Device: exercise training

INTERVENTIONS:
Device: exercise training — using either elastic band, dumbbells, treadmill, cycling, machines for 6 months

SUMMARY:
This study aimed to determine the ideal parameters of exercise program for frail middle-aged and older adults on physical and mental functions.

DETAILED DESCRIPTION:
Exercise has been suggested as a possible lifestyle intervention for improving physical and cognitive performance. Various training options depending on various physical circumstances will be presented. However, the ideal exercise protocol for frail middle-aged and older adults had the greater benefits remain unknown. In general, 3-6 months of frequent exercise can enhance physical and cognitive outcome.

The investigators conduct this multiple arm, prospective study to determine the ideal parameters of exercise program for frail middle-aged and older adults on physical and cognitive functions. This study designed to recruit 200 older adults with frailty. All the older adults will receive exercise training using either elastic band, dumbbells, machines, treadmill, cycling for 6 months. Outcome measures including a systematic evaluation for frail older persons using comprehensive geriatric assessment, as well as the assessments of physical and cognitive functions before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 50 years old with frailty syndrome

Exclusion Criteria:

* Acute illnesses, such as unstable cardiac dysrhythmia, sepsis, or unstable vital signs
* Physical or Cognitive issues that make it difficult for the patients to participate in our program

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of Barthel index | Up to 6 months
  Test function of activities of daily living, range from 0-100, higher values represent a greater outcome.
Change of Montreal Cognitive Assessment | Up to 6 months
  Test cognition including memory, attention, and language, range from 0-30, higher values represent a greater outcome
Change of Geriatric Depression Scale | Up to 6 months
  Test depression status, , range from 0-15, higher values represent a worse outcome
Change of Lawton Instrumental Activities of Daily Living (IADL) Scale | Up to 6 months
  To assesses a person's ability to perform tasks such as using a telephone, doing laundry, and handling finances.y. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent)

SECONDARY OUTCOMES:
Change of Six-minute Walking Test | Up to 6 months
  Test physical function. In healthy subjects, the 6-min walk distance ranges from 400 to 700 m.
Change of Timed Get-up-and-go Test | Up to 6 months
  Test for quantifying functional mobility
Change of Memory span test | Up to 6 months
  an examiner reads a list of random numbers aloud at about the rate of one number per second. At the end, the person being tested is asked to recall the items, in order.
Change of Color Trails Test | Up to 6 months
  Test cognitive function. Test is scored by how long it takes to complete the test.
Change of Digit symbol substitution test | Up to 6 months
  Test cognitive function. The test consists of filling as many empty boxes as possible with a symbol matching each number. The score is the number of correct number-symbol matches achieved.
Change of Mini-mental state examination | Up to 6 months
  Test cognitive function, range from 0-30, higher values represent a greater outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Sheng Lin, MD, Principal Investigator — Taipei Veterans General Hospital, Yuan-Shan/Su-Ao Branch, Yilan, Taiwan
Locations (1):
- Department of Physical Medicine & Rehabilitation, Taipei Veterans General Hospital, Yuan-Shan/Su-Ao Branch, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No